CLINICAL TRIAL: NCT03525847
Title: The Added Value of Contrast Enhancement for Guiding EUS-FNA in Solid Pancreatic Masses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Dr. Seicean Andrada (Other)
Responsible Party: Sponsor-Investigator, Professor Dr. Seicean Andrada, Principal Investigator Proffesor Dr Phd Md, Iuliu Hatieganu University of Medicine and Pharmacy
Organization: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 10430
Record Dates: First submitted 2017-11-16; First posted 2018-05-16 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Endoscopic Ultrasonography
Keywords: Contrast endosonograpy
MeSH Terms: interventions — Endosonography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- contrast enhanced FNA endosonography (Active Comparator): First passage in the solid pancreatic tumor using FNA endosonography then with the contrast enhanced FNA endosonography
  Interventions: Diagnostic Test: Endosonography
- FNA standard endosonography (Active Comparator): First passage in the solid pancreatic tumor using contrast enhanced FNA endosonography then with the FNA endosonography
  Interventions: Diagnostic Test: Endosonography

INTERVENTIONS:
Diagnostic Test: Endosonography — Puncture of the pancreatic solid mass with fine needle aspiration under endoscopic ultrasonographic control. Passage in the same pancreatic mass of first using standard FNA method then contrast enhanced FNA method or vice versa according to the randomization

SUMMARY:
A prospective study designed to show the superiority of contrast guided echoendoscopy versus conventional echoendoscopy

DETAILED DESCRIPTION:
A prospective study that compares the results using FNA contrast echoendoscopy versus standard FNA echoendoscopy in the diagnosis of solid pancreatic tumors

ELIGIBILITY:
Inclusion Criteria:

* solid pancreatic tumor lesions

Exclusion Criteria:

* severe coagulopathy of trombocytopenia <50.000
* patients refuse for biopsy prelevation or pacient's refuse to participate in the study

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CEUS FNA endosonography versus standard FNA endosonography in the etiological cyto histological of pancreatic solid tumors using histology core as comparison between the two methods | an average of 2 years
  Diagnostic accuracy of CEUS FNA endosonography versus standard FNA endosonography in the etiological cyto histological of pancreatic solid tumors using histology core as comparison between the two methods

SECONDARY OUTCOMES:
Quality of histological specimen(histology core) obtained with the two types of FNA biopsies (contrast enhanced and standard) | 5 days
  Visual analogic scale
Dysfunction in the two types of biopsies | day one
  failure or difficulty reports with each procedure (%)
Comparison between standand endosonography and contrast enhanced endosonography in obtaining a superior quality in obtaining histology core | day one
  Visual analogic scale

CONTACTS AND LOCATIONS:
Overall Officials: Seicean Andrada, Principal Investigator — Regional Institute of Gastroenterology and Hepatology "Octavian Fodor"Cluj-Napoca
Locations (1):
- Seicean Andrada, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No
The Study is used to show the superiority of CEUS-FNA endosonography Versus standard FNA endosonography in diagnosis of solid pancreatic masses

REFERENCES:
- [Background] Hou X, Jin Z, Xu C, Zhang M, Zhu J, Jiang F, Li Z. Contrast-enhanced harmonic endoscopic ultrasound-guided fine-needle aspiration in the diagnosis of solid pancreatic lesions: a retrospective study. PLoS One. 2015 Mar 20;10(3):e0121236. doi: 10.1371/journal.pone.0121236. eCollection 2015. PMID 25793739
- [Background] Yoshinaga S, Suzuki H, Oda I, Saito Y. Role of endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) for diagnosis of solid pancreatic masses. Dig Endosc. 2011 May;23 Suppl 1:29-33. doi: 10.1111/j.1443-1661.2011.01112.x. PMID 21535197
- [Result] Seicean A, Jinga M. Harmonic contrast-enhanced endoscopic ultrasound fine-needle aspiration: Fact or fiction? Endosc Ultrasound. 2017 Jan-Feb;6(1):31-36. doi: 10.4103/2303-9027.196917. PMID 28218198